CLINICAL TRIAL: NCT03749109
Title: A Randomised, Double-blind, Placebo-controlled, Proof-of-mechanism Phase 2 Trial Investigating the Effect of Quinagolide Extended-release Vaginal Ring on Reduction of Lesions Assessed by High-resolution Magnetic Resonance Imaging in Women With Endometrioma, Deep Infiltrating Endometriosis, and/or Adenomyosis
Brief Title: Quinagolide Vaginal Ring on Lesion Reduction Assessed by MRI in Women With Endometriosis/Adenomyosis
Acronym: QLARITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000295
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Endometriosis
Keywords: Endometrioma; Adenomyosis; Deep infiltrating endometriosis
MeSH Terms: conditions — Endometriosis; Adenomyosis | interventions — quinagolide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quinagolide 1080 µg (Experimental): Vaginal ring containing Quinagolide 1080 µg, with daily target release rate of 13.5 µg.
  Interventions: Drug: Quinagolide 1080 µg
- Placebo (Placebo Comparator): Vaginal ring containing matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinagolide 1080 µg — Vaginal ring containing Quinagolide 1080 µg for daily releases
  Other Names: FE 999051
  Arms: Quinagolide 1080 µg
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, proof-of-mechanism phase 2 trial investigating the effect of quinagolide extended-release vaginal ring on reduction of lesions assessed by high-resolution magnetic resonance imaging in women with endometrioma, deep infiltrating endometriosis, and/or adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal women between the ages 18-45 years (both inclusive) at the time of signing the informed consent
2. Body mass index (BMI) of 18-35 kg/m2 (both inclusive) at screening
3. Confirmation of deep infiltrating endometriosis (DIE), endometrioma or adenomyosis by high-resolution MRI at screening
4. Transvaginal ultrasound (TVU) documenting a uterus with no abnormalities of endometrium and presence of at least one ovary with no clinically significant abnormalities at screening. Note that presence of uterine fibroids are not exclusionary but presence of any submucosal fibroids or polyps are exclusionary
5. Willing and able to use a non-hormonal single-barrier method (i.e. condom) for contraception from the start of screening to the end-of-treatment. This is not required if adequate contraception is achieved by vasectomy of the male sexual partner, surgical sterilisation (e.g. tubal ligation and blockage methods such as ESSURE) of the subject, or true abstinence of the subject (sporadic sexual intercourse with men requiring condom use)
6. Willing to avoid the use of vaginal douches or any other intravaginally administered medications or devices (except for tampons) from randomization to the end of treatment

Exclusion Criteria:

1. Use of depot medroxyprogesterone acetate (MPA) within 10 months prior to the screening visit.
2. Use of gonadotropin-releasing (GnRH) agonists (3-month depot) or dopamine agonists within 6 months prior to the screening visit.
3. Use of GnRH agonists (1-month depot or nasal spray), GnRH antagonists, aromatase inhibitors, danazol, birth control implants (e.g. NEXPLANON), progestogen or levonorgestrel releasing intrauterine device (IUD) within 3 months prior to the screening visit.
4. Use of hormonal contraceptives (including combined oral contraceptive pill, transdermal patch, and contraceptive ring) within 1 menstrual cycle prior to the screening visit.
5. Contraindications to MRI such as having internal/external metallic devices and/or accessories (e.g. cardiac pacemakers and leg braces)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (11):
- Gyneacology Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Charité Universitätsmedizin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Münster, Münster
- Italy (4):
  - Azienda Opsedaliera Universitaria Careggi, Florence
  - Università degli Studi di Roma La Sapienza, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Poland (3):
  - Centrum Medyczne PROMED, Krakow
  - Gabinet Lekarski Specjalistyczny SONUS, Warsaw
  - Specjalistyczny Gabinet Lekarski, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellicer A, Taylor HS, Alberich-Bayarri A, Liu Y, Gamborg M, Barletta KE, Pinton P, Heiser PW, Bagger YZ. Quinagolide vaginal ring for reduction of endometriotic lesions: Results from the QLARITY trial. Eur J Obstet Gynecol Reprod Biol. 2025 Jun;310:113946. doi: 10.1016/j.ejogrb.2025.113946. Epub 2025 Mar 30. PMID 40188683

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed in 6 investigational sites in 3 countries between Aug 2019 to Jul 2021.
Pre-assignment Details: In total, 147 subjects were screened. Of these, 80 were screening failures and 67 were randomized and exposed to the investigational medicinal product (IMP): 35 to Quinagolide and 32 to Placebo.
Period: Overall Study
Arm/Group | Quinagolide 1080 µg | Placebo
Started | 35 | 32
Completed | 33 | 32
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quinagolide 1080 µg | Placebo | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 32 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (5.51) | 35.2 (5.96) | 36.1 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 32 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 32 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.91 (3.86) | 23.30 (4.15) | 23.62 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Sizes (mm) of Endometrioma, Deep Infiltrating Endometriosis (DIE) and Adenomyosis Lesions Summed by Type on Magnetic Resonance (MR) Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
  At screening, every measurable lesion (defined as ≥10 mm in size) of any type was recorded and was summed up by type for primary analysis.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: All analyses for primary and secondary efficacy endpoints are presented by lesion type. This means one subject can be included in multiple lesion groups, depending on the type of lesion(s) with a size of ≥10 mm present at baseline. Thus, the FAS population by lesion type includes 47 subjects in the endometrioma group, 45 subjects in the DIE group, and 36 subjects in the adenomyosis group. The primary and secondary efficacy results are presented for these subjects unless otherwise specified.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
mm
  Endometrioma: number analyzed (Participants) | 25 | 22
  Endometrioma | -0.20 (4.34) | -1.94 (4.48)
  DIE: number analyzed (Participants) | 19 | 26
  DIE | 2.41 (2.52) | -0.94 (2.03)
  Adenomyosis: number analyzed (Participants) | 20 | 16
  Adenomyosis | -3.10 (3.75) | -3.43 (3.87)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.78, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 1.74, 95% CI 2-sided [-10.45 to 13.94]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; DIE; Test type: Other; p = 0.29, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 3.35, 95% CI 2-sided [-2.89 to 9.59]
Statistical Analysis 3: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis; Test type: Other; p = 0.95, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.33, 95% CI 2-sided [-10.33 to 10.99]

2. Secondary Outcome: Percentage of Changes in the Sizes of Endometrioma, DIE and Adenomyosis Lesions Summed by Type on MR Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of changes in the size
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Percentage of changes in the size
  Endometrioma: number analyzed (Participants) | 22 | 21
  Endometrioma | 15.64 (70.12) | -6.83 (44.46)
  DIE: number analyzed (Participants) | 17 | 25
  DIE | 7.67 (15.22) | 5.81 (37.73)
  Adenomyosis: number analyzed (Participants) | 17 | 16
  Adenomyosis | -3.04 (32.31) | -6.99 (25.48)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.65, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -6.99, 95% CI 2-sided [-36.80 to 22.82]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; DIE; Test type: Other; p = 0.92, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -1.13, 95% CI 2-sided [-22.77 to 20.51]
Statistical Analysis 3: Comparison: Quinagolide 1080 µg vs Placebo; Test type: Other; p = 0.74, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -5.92, 95% CI 2-sided [-40.94 to 29.10]

3. Secondary Outcome: Proportion of Lesions by Type With a Decrease in a Size of ≥5 mm on MR Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Number analyzed (Lesions) | 112 | 108
Percentage of lesions
  Endometrioma: number analyzed (Lesions) | 53 | 46
  Endometrioma | 18.9 | 21.7
  DIE: number analyzed (Lesions) | 26 | 33
  DIE | 0 | 12.1
  Adenomyosis: number analyzed (Lesions) | 33 | 29
  Adenomyosis | 12.1 | 24.1
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.95, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.38 to 2.82]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis; Test type: Other; p = 0.39, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.14 to 2.17]

4. Secondary Outcome: Proportion of Subjects With a Lesion of Any Type Decreased in a Size of ≥5 mm on MR Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Percentage of subjects
  Endometrioma: number analyzed (Participants) | 25 | 22
  Endometrioma | 24.0 | 31.8
  DIE: number analyzed (Participants) | 19 | 26
  DIE | 0 | 11.5
  Adenomyosis: number analyzed (Participants) | 20 | 16
  Adenomyosis | 15.0 | 37.5
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.60, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.19 to 2.65]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis; Test type: Other; p = 0.21, Regression, Logistic; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.07 to 1.79]

5. Secondary Outcome: Number of New or Disappearing Endometrioma, DIE and Adenomyosis Lesions Summed by Type on MR Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: as for outcome 1
Measure: Number; unit: Lesions
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Lesions
  Endometrioma - Disappearing Lesions | 14 | 5
  DIE - Disappearing Lesions | 0 | 1
  Adenomyosis - Disappearing Lesions | 1 | 2
  Endometrioma - New Lesions | 3 | 3
  DIE - New Lesions | 0 | 0
  Adenomyosis - New Lesions | 0 | 0
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma - Disappearing Lesions; Test type: Other; p = 0.13, Negative-binomial regression; Rate Ratio = 2.53, 95% CI 2-sided [0.76 to 8.39]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis - Disappearing Lesions; Test type: Other; p = 0.56, Negative-binomial regression; Rate Ratio = 0.49, 95% CI 2-sided [0.04 to 5.41]

6. Secondary Outcome: Changes in the Volumes (mm3) of Endometrioma and DIE Lesions Summed by Type on MR Images at Cycle 4
Description: The MRI examination was performed on a high resolution 3T machine at screening and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: All analyses for primary and secondary efficacy endpoints are presented by lesion type. This means one subject can be included in multiple lesion groups, depending on the type of lesion(s) with a size of ≥10 mm present at baseline. Thus, the FAS population by lesion type includes 47 subjects in the endometrioma group, and 45 subjects in the DIE group. The primary and secondary efficacy results are presented for these subjects unless otherwise specified.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
mm^3
  Endometrioma: number analyzed (Participants) | 25 | 22
  Endometrioma | 2.12 (4.62) | 1.89 (4.77)
  DIE: number analyzed (Participants) | 19 | 26
  DIE | -0.15 (1.81) | -0.87 (1.25)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.97, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.23, 95% CI 2-sided [-12.78 to 13.23]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; DIE; Test type: Other; p = 0.74, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.72, 95% CI 2-sided [-3.63 to 5.07]

7. Secondary Outcome: Changes in the Sizes of Endometrioma Assessed by Transvaginal Ultrasound (TVU) at Cycle 4
Description: Transvaginal ultrasound (TVU) will be performed, preferably by the same sonographer, at the screening visit and at end-of-treatment / cycle 4.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 18 | 17
mm | 14.19 (8.70) | 4.06 (9.02)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Test type: Other; p = 0.42, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 10.13, 95% CI 2-sided [-14.74 to 35.00]

8. Secondary Outcome: Changes in the Mean Individual and Total Symptom and Sign Severity of Scores of the Biberoglu and Behrman (B&B) Scale at Cycle 4
Description: B&B scale is a used scale for endometriosis that consists of two parts, with the first part evaluating symptoms (i.e. different types of pain) and the second part evaluating physical signs.
  In the first part, the subject was asked to grade her pelvic pain (item A), dysmenorrhea (item B) and dyspareunia (item C) during the last menstrual cycle as none, mild, moderate or severe, corresponding to a score of 0-3.
  In the second part, the investigator graded the subject's pelvic tenderness (item D) and induration (item E) based on findings from a pelvic examination as none, mild, moderate or severe, corresponding to a score of 0-3.
  The total symptom and sign severity score was the sum of all five scores, i.e. A+B+C+D+E.
  The score can be between 0 and 15.
Time Frame: At baseline and at menstrual cycle 4 (around 4 months, each cycle is approximately 28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
score on a scale
  Endometrioma: number analyzed (Participants) | 24 | 22
  Endometrioma | -1.2 (2.26) | -2.1 (2.51)
  DIE: number analyzed (Participants) | 19 | 26
  DIE | -1.3 (2.16) | -1.6 (2.21)
  Adenomyosis: number analyzed (Participants) | 20 | 16
  Adenomyosis | -1.5 (2.33) | -1.9 (1.86)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma; Test type: Other; p = 0.10, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 1.09, 95% CI 2-sided [-0.20 to 2.38]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; DIE; Test type: Other; p = 0.67, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.28, 95% CI 2-sided [-1.02 to 1.58]
Statistical Analysis 3: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis; Test type: Other; p = 0.64, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.32, 95% CI 2-sided [-1.06 to 1.71]

9. Secondary Outcome: Changes in the Numerical Rating Scale (NRS) Pain Scores Per Cycle at Cycles 1, 2, 3 and 4
Description: Assessed by Subjects. NRS is a 11-point scale, with 0 indicating no pain and 10 indicating the worst imaginable pain.
  Subjects were asked to score the worst pain in relation to endometriosis / adenomyosis on the NRS based on a recall of their experiences during the following timeframes:
  * during the last menstrual cycle
  * during the menstrual period of the last menstrual cycle
  * during the non-menstrual period of the last menstrual cycle
Time Frame: At baseline and at menstrual cycles 1 (~1 month), 2 (~2 months), 3 (~3 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
score on a scale
  Endometrioma at cycle 1: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 1 | -0.5 (1.96) | -0.7 (2.21)
  Endometrioma at cycle 2: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 2 | -0.9 (2.17) | -1.1 (2.85)
  Endometrioma at cycle 3: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 3 | -1.7 (2.73) | -1.1 (1.67)
  Endometrioma at cycle 4: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 4 | -1.5 (3.11) | -2.0 (1.94)
  DIE at cycle 1: number analyzed (Participants) | 19 | 26
  DIE at cycle 1 | -0.6 (2.14) | -0.7 (2.19)
  DIE at cycle 2: number analyzed (Participants) | 19 | 26
  DIE at cycle 2 | -1.1 (2.20) | -1.4 (2.97)
  DIE at cycle 3: number analyzed (Participants) | 19 | 26
  DIE at cycle 3 | -1.7 (2.65) | -1.0 (1.97)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | -1.2 (2.27) | -2.1 (2.21)
  Adenomyosis at cycle 1: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 1 | 0.3 (1.84) | -0.7 (2.24)
  Adenomyosis at cycle 2: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 2 | -0.7 (2.37) | -0.9 (2.13)
  Adenomyosis at cycle 3: number analyzed (Participants) | 19 | 16
  Adenomyosis at cycle 3 | -0.8 (2.34) | -0.9 (1.78)
  Adenomyosis at cycle 4: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 4 | -1.6 (2.91) | -1.9 (2.28)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 1; Test type: Other; p = 0.73, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.21, 95% CI 2-sided [-1.02 to 1.44]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 2; Test type: Other; p = 0.54, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.42, 95% CI 2-sided [-0.97 to 1.82]
Statistical Analysis 3: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 3; Test type: Other; p = 0.46, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -0.50, 95% CI 2-sided [-1.86 to 0.85]
Statistical Analysis 4: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 4; Test type: Other; p = 0.49, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.53, 95% CI 2-sided [-0.99 to 2.05]
Statistical Analysis 5: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 1; Test type: Other; p = 0.99, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -0.01, 95% CI 2-sided [-1.32 to 1.30]
Statistical Analysis 6: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 2; Test type: Other; p = 0.83, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.17, 95% CI 2-sided [-1.38 to 1.71]
Statistical Analysis 7: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 3; Test type: Other; p = 0.28, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -0.74, 95% CI 2-sided [-2.11 to 0.63]
Statistical Analysis 8: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 4; Test type: Other; p = 0.26, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.75, 95% CI 2-sided [-0.57 to 2.07]
Statistical Analysis 9: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 1; Test type: Other; p = 0.19, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.91, 95% CI 2-sided [-0.49 to 2.31]
Statistical Analysis 10: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 2; Test type: Other; p = 0.93, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.07, 95% CI 2-sided [-1.45 to 1.58]
Statistical Analysis 11: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 3; Test type: Other; p = 0.85, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -0.13, 95% CI 2-sided [-1.58 to 1.32]
Statistical Analysis 12: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 4; Test type: Other; p = 0.99, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 0.01, 95% CI 2-sided [-1.68 to 1.69]

10. Secondary Outcome: Changes in the Endometriosis Health Profile-30 (EHP-30) Scores at Cycles 2 and 4
Description: EHP-30 is a quality-of-life questionnaire. Score ranges from 0-100 and lower score denotes improvement.
  It consists of 30 questions measuring the frequency of the endometriosis impact on their quality of life during the past four weeks, with five options of never, rarely, sometimes, often and always.
Time Frame: At baseline, at menstrual cycles 2 (~2 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Score on a scale
  Endometrioma at cycle 2: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 2 | -46.6 (90.49) | -51.0 (71.60)
  Endometrioma at cycle 4: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 4 | -56.6 (88.84) | -94.0 (85.14)
  DIE at cycle 2: number analyzed (Participants) | 19 | 26
  DIE at cycle 2 | -55.6 (91.14) | -41.7 (86.27)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | -54.8 (87.29) | -85.7 (98.96)
  Adenomyosis at cycle 2: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 2 | -46.3 (102.92) | -33.2 (52.21)
  Adenomyosis at cycle 4: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 4 | -64.9 (105.62) | -79.4 (90.04)
Statistical Analysis 1: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 2; Test type: Other; p = 0.75, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -7.35, 95% CI 2-sided [-53.97 to 39.27]
Statistical Analysis 2: Comparison: Quinagolide 1080 µg vs Placebo; Endometrioma at cycle 4; Test type: Other; p = 0.42, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 17.31, 95% CI 2-sided [-25.41 to 60.04]
Statistical Analysis 3: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 2; Test type: Other; p = 0.47, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -17.66, 95% CI 2-sided [-66.30 to 30.98]
Statistical Analysis 4: Comparison: Quinagolide 1080 µg vs Placebo; DIE at cycle 4; Test type: Other; p = 0.27, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 25.61, 95% CI 2-sided [-21.05 to 72.27]
Statistical Analysis 5: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 2; Test type: Other; p = 0.41, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = -20.95, 95% CI 2-sided [-71.83 to 29.92]
Statistical Analysis 6: Comparison: Quinagolide 1080 µg vs Placebo; Adenomyosis at cycle 4; Test type: Other; p = 0.93, ANCOVA; ANCOVA adjusted for baseline lesion size; Difference in LS mean = 2.25, 95% CI 2-sided [-49.57 to 54.06]

11. Secondary Outcome: Changes in the Menstrual Bleeding Pattern Over 4 Cycles (Menstrual Cycle Duration)
Description: Assessed by subject self-reported answers to menstrual bleeding questions. The Menstrual Cycle Duration is shown.
Time Frame: At baseline and at menstrual cycles 1 (~1 month), 2 (~2 months), 3 (~3 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Days
  Endometrioma at baseline: number analyzed (Participants) | 25 | 22
  Endometrioma at baseline | 31.9 (10.54) | 32.6 (10.38)
  Endometrioma at cycle 1: number analyzed (Participants) | 23 | 22
  Endometrioma at cycle 1 | 27.8 (2.92) | 26.9 (2.39)
  Endometrioma at cycle 2: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 2 | 28.1 (2.13) | 27.4 (2.50)
  Endometrioma at cycle 3: number analyzed (Participants) | 22 | 23
  Endometrioma at cycle 3 | 27.7 (2.12) | 28.3 (2.65)
  Endometrioma at cycle 4: number analyzed (Participants) | 23 | 23
  Endometrioma at cycle 4 | 28.2 (3.27) | 26.9 (2.23)
  DIE at baseline: number analyzed (Participants) | 19 | 26
  DIE at baseline | 33.2 (11.80) | 31.4 (9.45)
  DIE at cycle 1: number analyzed (Participants) | 18 | 26
  DIE at cycle 1 | 26.7 (2.66) | 27.3 (2.78)
  DIE at cycle 2: number analyzed (Participants) | 18 | 26
  DIE at cycle 2 | 27.4 (1.98) | 27.7 (2.52)
  DIE at cycle 3: number analyzed (Participants) | 17 | 27
  DIE at cycle 3 | 28.2 (2.86) | 28.5 (2.29)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | 26.9 (2.23) | 27.7 (2.59)
  Adenomyosis at baseline: number analyzed (Participants) | 20 | 16
  Adenomyosis at baseline | 33.5 (11.16) | 32.4 (11.49)
  Adenomyosis at cycle 1: number analyzed (Participants) | 19 | 16
  Adenomyosis at cycle 1 | 27.7 (2.54) | 26.8 (2.61)
  Adenomyosis at cycle 2: number analyzed (Participants) | 19 | 16
  Adenomyosis at cycle 2 | 28.3 (2.23) | 27.4 (2.37)
  Adenomyosis at cycle 3: number analyzed (Participants) | 16 | 17
  Adenomyosis at cycle 3 | 27.8 (2.52) | 27.9 (1.93)
  Adenomyosis at cycle 4: number analyzed (Participants) | 18 | 17
  Adenomyosis at cycle 4 | 27.2 (1.50) | 27.4 (1.87)

12. Secondary Outcome: Changes in the Menstrual Bleeding Pattern Over 4 Cycles (Menstrual Bleeding Duration)
Description: Assessed by subject self-reported answers to menstrual bleeding questions. The Menstrual Bleeding Duration is shown.
Time Frame: At baseline and at menstrual cycles 1 (~1 month), 2 (~2 months), 3 (~3 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Days
  Endometrioma at baseline: number analyzed (Participants) | 25 | 22
  Endometrioma at baseline | 5.1 (1.08) | 5.1 (0.97)
  Endometrioma at cycle 1: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 1 | 5.3 (1.71) | 4.7 (0.77)
  Endometrioma at cycle 2: number analyzed (Participants) | 25 | 22
  Endometrioma at cycle 2 | 5.3 (1.22) | 5.1 (0.87)
  Endometrioma at cycle 3: number analyzed (Participants) | 24 | 23
  Endometrioma at cycle 3 | 4.5 (1.61) | 4.8 (0.89)
  Endometrioma at cycle 4: number analyzed (Participants) | 26 | 24
  Endometrioma at cycle 4 | 5.0 (1.43) | 4.7 (1.52)
  DIE at baseline: number analyzed (Participants) | 19 | 26
  DIE at baseline | 4.9 (0.99) | 5.3 (1.01)
  DIE at cycle 1: number analyzed (Participants) | 19 | 26
  DIE at cycle 1 | 5.0 (1.60) | 4.6 (0.70)
  DIE at cycle 2: number analyzed (Participants) | 20 | 26
  DIE at cycle 2 | 5.0 (1.82) | 5.0 (1.04)
  DIE at cycle 3: number analyzed (Participants) | 19 | 27
  DIE at cycle 3 | 4.5 (1.22) | 4.9 (0.93)
  DIE at cycle 4: number analyzed (Participants) | 20 | 27
  DIE at cycle 4 | 5.2 (1.04) | 4.9 (1.60)
  Adenomyosis at baseline: number analyzed (Participants) | 20 | 16
  Adenomyosis at baseline | 5.2 (1.20) | 5.4 (1.15)
  Adenomyosis at cycle 1: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 1 | 5.0 (1.75) | 4.9 (0.62)
  Adenomyosis at cycle 2: number analyzed (Participants) | 21 | 16
  Adenomyosis at cycle 2 | 4.6 (1.78) | 4.8 (1.17)
  Adenomyosis at cycle 3: number analyzed (Participants) | 19 | 17
  Adenomyosis at cycle 3 | 4.3 (1.66) | 4.7 (1.05)
  Adenomyosis at cycle 4: number analyzed (Participants) | 21 | 17
  Adenomyosis at cycle 4 | 5.0 (0.74) | 5.0 (1.32)

13. Secondary Outcome: Serum Levels of Prolactin During Cycle 1, at Cycles 2 and 4
Description: Assessed by blood sample collection
Time Frame: Within 1-5 days post randomization, and at menstrual cycles 2 (~2 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
pg/L
  Endometrioma at cycle 1: number analyzed (Participants) | 24 | 21
  Endometrioma at cycle 1 | 5.51 (3.604) | 12.68 (4.618)
  Endometrioma at cycle 2: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 2 | 9.30 (4.739) | 12.79 (4.381)
  Endometrioma at cycle 4: number analyzed (Participants) | 25 | 22
  Endometrioma at cycle 4 | 9.47 (4.081) | 12.31 (6.648)
  DIE at cycle 1: number analyzed (Participants) | 19 | 25
  DIE at cycle 1 | 5.95 (3.258) | 10.80 (4.201)
  DIE at cycle 2: number analyzed (Participants) | 19 | 26
  DIE at cycle 2 | 10.36 (5.118) | 11.85 (5.029)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | 10.65 (4.465) | 12.08 (6.739)
  Adenomyosis at cycle 1: number analyzed (Participants) | 20 | 15
  Adenomyosis at cycle 1 | 5.80 (4.017) | 12.13 (4.563)
  Adenomyosis at cycle 2: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 2 | 7.97 (2.608) | 11.94 (4.150)
  Adenomyosis at cycle 4: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 4 | 9.35 (3.418) | 11.95 (4.395)

14. Secondary Outcome: Serum Levels of Thyroid-stimulating Hormone (TSH) During Cycle 1, at Cycles 2 and 4
Description: Assessed by blood sample collection
Time Frame: Within 1-5 days post randomization, and at menstrual cycles 2 (~2 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
mIU/L
  Endometrioma at cycle 1: number analyzed (Participants) | 24 | 21
  Endometrioma at cycle 1 | 1.672 (1.3376) | 1.513 (0.6822)
  Endometrioma at cycle 2: number analyzed (Participants) | 24 | 22
  Endometrioma at cycle 2 | 1.785 (1.0535) | 1.509 (0.6746)
  Endometrioma at cycle 4: number analyzed (Participants) | 25 | 22
  Endometrioma at cycle 4 | 1.692 (0.9489) | 1.422 (0.6528)
  DIE at cycle 1: number analyzed (Participants) | 19 | 25
  DIE at cycle 1 | 1.706 (1.5550) | 1.394 (0.8200)
  DIE at cycle 2: number analyzed (Participants) | 19 | 26
  DIE at cycle 2 | 1.726 (1.1633) | 1.383 (0.6903)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | 1.375 (0.8953) | 1.299 (0.6571)
  Adenomyosis at cycle 1: number analyzed (Participants) | 20 | 15
  Adenomyosis at cycle 1 | 2.067 (1.8100) | 1.325 (0.7248)
  Adenomyosis at cycle 2: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 2 | 1.722 (1.1557) | 1.311 (0.5664)
  Adenomyosis at cycle 4: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 4 | 1.801 (0.9463) | 1.353 (0.5614)

15. Secondary Outcome: Serum Levels of Insulin-like Growth Factor-1 (IGF-1) During Cycle 1, at Cycles 2 and 4
Description: Assessed by blood sample collection
Time Frame: Within 1-5 days post randomization, and at menstrual cycles 2 (~2 months) and 4 (~4 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
nmol/L
  Endometrioma at cycle 1: number analyzed (Participants) | 24 | 21
  Endometrioma at cycle 1 | 23.90 (8.002) | 22.96 (6.721)
  Endometrioma at cycle 2: number analyzed (Participants) | 23 | 22
  Endometrioma at cycle 2 | 19.9 (6.511) | 21.81 (5.481)
  Endometrioma at cycle 4: number analyzed (Participants) | 25 | 22
  Endometrioma at cycle 4 | 21.82 (5.450) | 20.22 (5.786)
  DIE at cycle 1: number analyzed (Participants) | 19 | 25
  DIE at cycle 1 | 22.16 (8.099) | 23.68 (6.135)
  DIE at cycle 2: number analyzed (Participants) | 19 | 26
  DIE at cycle 2 | 18.01 (5.484) | 21.07 (6.526)
  DIE at cycle 4: number analyzed (Participants) | 19 | 26
  DIE at cycle 4 | 20.98 (5.678) | 20.53 (6.083)
  Adenomyosis at cycle 1: number analyzed (Participants) | 20 | 15
  Adenomyosis at cycle 1 | 21.80 (7.763) | 22.51 (4.580)
  Adenomyosis at cycle 2: number analyzed (Participants) | 19 | 16
  Adenomyosis at cycle 2 | 19.17 (6.497) | 19.93 (5.233)
  Adenomyosis at cycle 4: number analyzed (Participants) | 20 | 16
  Adenomyosis at cycle 4 | 21.19 (6.331) | 18.93 (4.836)

16. Secondary Outcome: Plasma Concentrations of Quinagolide and Its Metabolites During Cycles 1 to 4
Description: Assessed by blood sample collection
Time Frame: Within 1-5 days post randomization, within 7-14 days post randomization, and at menstrual cycles 1 (~1 month), 2 (~2 months), 3 (~3 months) and 4 (~4 months)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Quinagolide 1080 μg: Vaginal ring containing Quinagolide 1080 μg, with daily target release rate of 13.5 μg.
  Quinagolide 1080 μg: Vaginal ring containing Quinagolide 1080 μg for daily releases
Arm/Group | Quinagolide 1080 μg
Number analyzed (Participants) | 33
pg/mL
  Within 1-5 days of randomization: number analyzed (Participants) | 30
  Within 1-5 days of randomization | 11.66 (5.23)
  Within 7-14 days of randomization: number analyzed (Participants) | 32
  Within 7-14 days of randomization | 5.50 (2.59)
  Cycle 1: number analyzed (Participants) | 32
  Cycle 1 | 2.90 (1.33)
  Cycle 2 | 2.92 (1.68)
  Cycle 3: number analyzed (Participants) | 32
  Cycle 3 | 2.78 (1.32)
  Cycle 4: number analyzed (Participants) | 32
  Cycle 4 | 3.16 (3.03)

17. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Hematocrit
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: % v/v
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 33 | 32
% v/v | -0.007 (0.0181) | -0.005 (0.0259)

18. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Hemaglobin
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 34 | 32
g/L | -3.6 (5.60) | -3.2 (8.69)

19. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Ery. Mean Corpuscular Hemoglobin
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 34 | 32
pg/cell | -0.7 (0.71) | -0.6 (1.22)

20. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Ery. Mean Corpuscular HGB Concentration
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 33 | 32
g/L | -3.1 (7.11) | -4.3 (8.76)

21. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Ery. Mean Corpuscular Volume
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 33 | 32
fL | -1.2 (2.11) | -0.7 (3.10)

22. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Platelets
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 34 | 31
10^9 cells/L | 4.9 (33.98) | 11.6 (45.92)

23. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Erythrocytes
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 34 | 32
10^12 cells/L | -0.02 (0.192) | -0.01 (0.228)

24. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Leukocytes
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 34 | 32
10^9 cells/L | -0.43 (1.928) | 0.18 (2.055)

25. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Alanine Aminotransferase
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
U/L | -1.1 (5.88) | -0.2 (3.86)

26. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Albumin
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
g/L | 0.0 (2.28) | 0.7 (2.84)

27. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Alkaline Phosphatase
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
IU/L | 3.1 (8.18) | 4.2 (6.67)

28. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Aspartate Aminotransferase
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
U/L | 1.0 (3.72) | 0.5 (3.43)

29. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Bicarbonate
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | -2.7 (2.59) | -2.9 (2.51)

30. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Direct Bilirubin
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
umol/L | 0.0 (0.38) | 0.0 (1.10)

31. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Bilirubin
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
umol/L | -1.2 (2.84) | -0.8 (4.57)

32. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Calcium
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | 0.009 (0.0896) | 0.012 (0.0773)

33. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Chloride
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | 0.2 (2.68) | -0.5 (2.49)

34. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Cholesterol
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | 0.045 (0.5050) | 0.244 (0.5219)

35. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Creatinine
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
umol/L | -3.5 (8.21) | -4.3 (7.82)

36. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Gamma Glutamyl Transferase
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
U/L | -1.1 (4.77) | 1.0 (4.46)

37. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Glucose
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | -0.07 (0.734) | -0.06 (0.866)

38. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Lactate Dehydrogenase
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
U/L | 2.7 (12.30) | 2.8 (8.42)

39. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Phosphate
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | -0.013 (0.1452) | 0.048 (0.1885)

40. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Potassium
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | 0.07 (0.333) | 0.06 (0.357)

41. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Sodium
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | 0.7 (2.04) | 0.4 (2.54)

42. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Protein
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
g/L | -0.1 (3.82) | 1.4 (3.19)

43. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Urate
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
umol/L | 10.7 (56.36) | 1.3 (37.59)

44. Secondary Outcome: Changes in Clinical Chemistry and Hematology Parameters: Urea Nitrogen
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Population: Subjects analyzed for this endpoint represent subjects who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 31
mmol/L | -0.180 (1.0184) | 0.148 (1.2286)

45. Secondary Outcome: Proportion of Subjects With Markedly Abnormal Changes in Clinical Chemistry and Hematology Parameters
Description: Assessed by blood sample collection
Time Frame: At baseline and at menstrual cycle 4 (around 5 months, each cycle is approximately 28 days)
Measure: Number; unit: Percentage of subjects
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Percentage of subjects | 2.86 | 0

46. Secondary Outcome: Frequency and Intensity of Adverse Events
Description: Assessed by and Adverse Event Log completed by the Investigator
Time Frame: From obtaining the informed consent to end of trial (up to 6 menstrual cycles ~ around 6 months, each cycle is approximately 28 days)
Measure: Number; unit: Percentage of subjects
Arm/Group | Quinagolide 1080 µg | Placebo
Number analyzed (Participants) | 35 | 32
Percentage of subjects
  Mild adverse events | 28.6 | 43.8
  Moderate adverse events | 42.9 | 37.5
  Severe adverse events | 2.9 | 9.4

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each participant from the time of signed informed consent for participation in the trial to follow-up visit (approximately 1 month after visit 8 (month 4), up to 5 months).
Description: All adverse events with onset after start of first administration of IMP and before the follow-up phone call were considered treatment-emergent.
Arm/Group | Quinagolide 1080 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/32
Other Adverse Events (participants affected / at risk) | 20/35 | 20/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinagolide 1080 µg (N=35) | Placebo (N=32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinagolide 1080 µg (N=35) | Placebo (N=32)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (4)
Fatigue (General disorders) | 1 (1) | 2 (2)
Peripheral swelling (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 6 (9) | 8 (15)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 2 (4) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03749109/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03749109/SAP_001.pdf